CLINICAL TRIAL: NCT00784589
Title: Comparison Between Monoclonal Antibody CD20 Treatment (Rituximab (mabthéra))and General Corticotherapy Treatment in Patients With Pemphigus
Brief Title: Comparison Between Rituximab Treatment and General Corticotherapy Treatment in Patients With Pemphigus
Acronym: Rituximab 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008/068/HP
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Pemphigus Disease
Keywords: Corticothérapy; Rituximab; therapeutic efficacity; therapeutic tolerance
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Experimental)
  Interventions: Drug: Rituximab
- Corticotherapy (Active Comparator): General Corticotherapy
  Interventions: Drug: General Corticotherapy

INTERVENTIONS:
Drug: General Corticotherapy — for patients with severe pemphigus : general corticotherapy Arm : 1.5mg/kg/d for 1 month, then 1.25mg/kg/d for 1 month, then 1mg/kg/d for 1 month, then 0.75 mg/kg/d for 1 month, then 0.5 mg/kg/d for 3 months, then 0.3 mg/kg/d for 3 months, then 0.2 mg/kg/d for 4 months, then 0.1 mg/kg/d for 4 months, for patients with moderated pemphigus : general corticotherapy Arm : 1mg/kg/d for 1 month, then 0.75mg/kg/d for 1 month, then 0.5mg/kg/d for 2 months, then 0.3 mg/kg/d for 2 months, then 0.2 mg/kg/d for 3 months, then 0.1 mg/kg/d for 3 months,
  Arms: Corticotherapy
Drug: Rituximab — for patients with severe pemphigus : rituximab Arm : 1mg/kg/d for 1 month, then 0.75 mg/kg/d for 1 month, then 0.5 mg/kg/d for 1 month, then 0.3 mg/kg/d for 1 month, then 0.2 mg/kg/d for 1 month, then 0.1 mg/kg/d for 1 month for patients with moderated pemphigus : rituximab Arm : 0.5mg/kg/d for 1 month, then 0.30 mg/kg/d for 1 month, then 0.2 mg/kg/d for 1 month,
  Arms: Rituximab

SUMMARY:
Pemphigus is a severe and sometimes life-threatening disease with a mortality rate between 5 and 10 percent depending on the severity of disease and age of patients.

The standard of care is high doses of corticosteroids (CS) (usually, prednisone, 1 to 1.5. mg/kg/day, which are often associated with immunosuppressive drugs i.e., azathioprine, mycophenolate mofetil, cyclophosphamide, cyclosporine, although only one randomised study has demonstrated the superiority of the combination of corticosteroids and immunosuppressive drugs as compared to corticosteroids alone (9). Because of the low frequency of the disease, control trials are difficult to conduct. Evaluation of the different treatment regimens proposed, i;e; corticosteroids alone, CS and immunosuppressive drugs, IV immunoglobulins or new therapeutic regimens such as rituximab (an anti-CD20 monoclonal antibody directed against B- lymphocytes) or immunoadsorbtion.

ELIGIBILITY:
Inclusion Criteria:

* age >=18 and <= 80years
* consent obtained from patient
* effective female contraceptive method for women in procreate age
* new case of pemphigus vulgaris (PV) or pemphigus foliaceus (PF)

Exclusion Criteria:

* pemphigus vulgaris (PV) or pemphigus foliaceus (PF) treated
* pregnant woman or nursing mother
* woman able to have a baby and without contraception during the clinical trial period
* age < 18 or > 80
* karnovsky < 50%
* serious antecedents of allergy or anaphylactic reaction with human monoclonal antibody
* patient with depletion lymphocytic treatment in the next month
* unstable angina or ischemic heart disease
* cardiac insufficiency
* cardiac rhythm trouble uncontrolled
* positive HIV serology
* positive hepatitis B and / or C serology
* no consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-07; Primary Completion 2013-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with pemphigus controlled 24 months after the start of Rituximab treatment | 2 years

SECONDARY OUTCOMES:
Number of patients with pemphigus with both cutaneous and mucosal lesions healing after 6 months of rituximab treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pascal JOLY, Professor, Principal Investigator — Clinique Dermatologique - Hôpitaux de Rouen
Locations (1):
- CHU de Rouen - Hôpitaux de Rouen, Rouen, Seine Maritime, France

REFERENCES:
- [Derived] Mignard C, Maho-Vaillant M, Golinski ML, Balaye P, Prost-Squarcioni C, Houivet E, Calbo SB, Labeille B, Picard-Dahan C, Konstantinou MP, Chaby G, Richard MA, Bouaziz JD, Duvert-Lehembre S, Delaporte E, Bernard P, Caux F, Alexandre M, Ingen-Housz-Oro S, Vabres P, Quereux G, Dupuy A, Debarbieux S, Avenel-Audran M, D'Incan M, Bedane C, Beneton N, Jullien D, Dupin N, Misery L, Machet L, Beylot-Barry M, Dereure O, Sassolas B, Benichou J, Joly P, Hebert V; French Study Group on Autoimmune Bullous Skin Diseases. Factors Associated With Short-term Relapse in Patients With Pemphigus Who Receive Rituximab as First-line Therapy: A Post Hoc Analysis of a Randomized Clinical Trial. JAMA Dermatol. 2020 May 1;156(5):545-552. doi: 10.1001/jamadermatol.2020.0290. PMID 32186656
- [Derived] Joly P, Maho-Vaillant M, Prost-Squarcioni C, Hebert V, Houivet E, Calbo S, Caillot F, Golinski ML, Labeille B, Picard-Dahan C, Paul C, Richard MA, Bouaziz JD, Duvert-Lehembre S, Bernard P, Caux F, Alexandre M, Ingen-Housz-Oro S, Vabres P, Delaporte E, Quereux G, Dupuy A, Debarbieux S, Avenel-Audran M, D'Incan M, Bedane C, Beneton N, Jullien D, Dupin N, Misery L, Machet L, Beylot-Barry M, Dereure O, Sassolas B, Vermeulin T, Benichou J, Musette P; French study group on autoimmune bullous skin diseases. First-line rituximab combined with short-term prednisone versus prednisone alone for the treatment of pemphigus (Ritux 3): a prospective, multicentre, parallel-group, open-label randomised trial. Lancet. 2017 May 20;389(10083):2031-2040. doi: 10.1016/S0140-6736(17)30070-3. Epub 2017 Mar 22. PMID 28342637